CLINICAL TRIAL: NCT02181426
Title: Dose Response of Ketorolac in Out-Patients Undergoing Knee Arthroscopy
Brief Title: Dose Response of Ketorolac in Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ketorolac Knee Arthroscopy
Record Dates: First submitted 2014-06-26; First posted 2014-07-04 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Meniscectomy
Keywords: Knee Arthroscopy
MeSH Terms: interventions — Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0 mg of Ketorolac (Placebo Comparator): participant receives 0 mg of Ketorolac
  Interventions: Drug: Ketorolac Dose
- 7.5 mg of Ketorolac (Active Comparator): participant receives 7.5 mg of Ketorolac
  Interventions: Drug: Ketorolac Dose
- 15 mg Ketorolac (Active Comparator): participant receives 15 mg of Ketorolac
  Interventions: Drug: Ketorolac Dose
- 30 mg Ketorolac (Active Comparator): participant receives 30mg of Ketorolac
  Interventions: Drug: Ketorolac Dose

INTERVENTIONS:
Drug: Ketorolac Dose — Subjects will be assigned an enrollment number. Enrollment numbers will be assigned consecutively in the order of study enrollment. Based on the enrollment number, subjects will be randomized by a pre-determined computer randomization list created by a statistician to receive a ketorolac dose (0, 7.5, 15, 30 mg).
  Other Names: Toradol

SUMMARY:
Ketorolac is administered as current practice to the majority of patients undergoing knee arthroscopy, the appropriate dose of ketorolac to be administered has not been evaluated.

DETAILED DESCRIPTION:
Past studies have examined different doses of ketorolac administered to patients after spinal fusion surgery and found that 7.5 mg every 6 hours was as effective as 15 or 30 mg every 6 hours in decreasing postoperative pain and patient opiate consumption. Since ketorolac side effects such as gastrointestinal and surgical site bleeding seem to be dose related, utilizing a lower dose of ketorolac may be more efficacious.

ELIGIBILITY:
Population: Patients scheduled for outpatient knee arthroscopy under general anesthesia with ASA physical status I-III ages 18-65 years old. All subjects will receive informed consent. Subjects will not be eligible to participate if they cannot provide informed consent. Non-English speaking patients will not be included due to the limited time and availability of translators.

Inclusion Criteria:

1. Ability to consent and desire to participate in study
2. Outpatient knee arthroscopy with Dr. C. David Geier
3. ASA physical status I-III
4. 18-65 years old
5. Over 50 kg (110 pounds)
6. General anesthesia

Exclusion Criteria

1. Any contraindication to receiving a non-steroidal antiinflammatory medication (including but not limited to allergy to any non-steroidal antiinflammatory medications including aspirin; chronic renal insufficiency; history of gastric ulcers, gastritis, peptic ulcers or gastrointestinal bleeding; severe volume depletion; presence of cerebrovascular bleeding or high risk of bleeding)
2. Allergy to propofol, fentanyl or hydromorphone.
3. Any chronic painful conditions requiring opioid use for over the last 6 months
4. Emergency surgery
5. Altered mental status (not oriented to place, person or time)
6. Pregnant or lactating patients
7. Patient is taking non-steroidal antiinflammatory medications (including aspirin)1 at home and took that medication on day of surgery.
8. Non-English speaking
9. Patient refusal to study
10. Patient refusal or not a candidate for general anesthesia with Laryngeal Mask Airway (LMA)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-03; Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia H Wilson, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0 mg of Ketorolac | 7.5 mg of Ketorolac | 15 mg Ketorolac | 30 mg Ketorolac
Started | 28 | 28 | 28 | 28
Completed | 28 | 28 | 28 | 28
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0 mg of Ketorolac | 7.5 mg of Ketorolac | 15 mg Ketorolac | 30 mg Ketorolac | Total
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 112
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 28 | 28 | 112
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.4 (11.9) | 44.2 (12.7) | 44.7 (14.2) | 44.4 (13) | 45.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 15 | 12 | 49
  Male | 14 | 20 | 13 | 16 | 63
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 28 | 28 | 28 | 112

OUTCOME MEASURES:

1. Primary Outcome: PACU Opiate Consumption
Description: Total PACU opioid consumption measured in intravenous morphine mg equivalents (IV MME).
Time Frame: Less than 1 day (PACU stay in the postoperative period)
Population: The study enrolled 112 patient with 28 patients randomized to each group.
Measure: Mean (Standard Error); unit: IV Morphine Equivalents (mg)
Arm/Group | 0 mg of Ketorolac | 7.5 mg of Ketorolac | 15 mg Ketorolac | 30 mg Ketorolac
Number analyzed (Participants) | 28 | 28 | 28 | 28
IV Morphine Equivalents (mg) | 7.7 (0.86) | 6.3 (0.86) | 6.5 (0.86) | 5.0 (0.86)

ADVERSE EVENTS:
Arm/Group | 0 mg of Ketorolac | 7.5 mg of Ketorolac | 15 mg Ketorolac | 30 mg Ketorolac
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No